CLINICAL TRIAL: NCT03097796
Title: An Open-Label, Multiple Ascending Dose Study to Evaluate the Safety and Tolerability of PUL-042 Inhalation Solution in Subjects With Hematologic Malignancies and Recipients of Stem Cell Transplantation
Brief Title: A Multiple Ascending Dose Study of PUL-042 in Stem Cell Transplant Recipients
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Development plan revised
Sponsor: Pulmotect, Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PUL-042-201A; R44HL127677 (NIH)
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Hematologic Diseases; Stem Cell Transplants
MeSH Terms: conditions — Hematologic Diseases | interventions — Pam2CSK4 acetate and ODN M362 combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PUL-042 (Experimental): PUL-042 Inhalation Solution
  Interventions: Drug: PUL-042

INTERVENTIONS:
Drug: PUL-042 — PUL-042 Inhalation Solution

SUMMARY:
Subjects with hematologic malignancies or recipients of a first allogenic or autologus hematopoietic stem cell transplant, without any evidence or respiratory infection, will receive 4 doses of PUL-042 Inhalation Solution over a 2 week period. Subjects will be evaluated for tolerability of the drug. If tolerated, dose escalation may occur with up to 4 dose levels tested

DETAILED DESCRIPTION:
This is an open-label multiple ascending dose study with a 3+3 study design to examine the safety and tolerability of PUL-042 Inhalation Solution in subjects with hematologic malignancies or recipients of a first allogenic or autologus hematopoietic stem cell transplant. Subjects will receive 4 doses over 2 weeks.

Cohort size will be 3 subjects, once 3 subjects have completed treatment and follow-up at a dose level, subject data will be evaluated by an independent data safety monitoring committee prior to dosing additional subjects. The Committee may recommend increasing the dose, maintaining the same dose, or decreasing the dose.

Once the maximum dose is determined, there may be up to 6 additional subjects dosed at that level.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with hematologic malignancies or recipients of a first allogeneic or autologous hematopoietic stem cell transplantation and presently clinically stable
2. Pulse oximetry of hemoglobin saturation ≥92% on room air
3. Adult (≥18 years)
4. Spirometry (FEV1 and forced vital capacity [FVC]) ≥80% of predicted value
5. If female, must be either post-menopausal (one year or greater without menses), surgically sterile, or, for female subjects of child-bearing potential who are capable of conception must be: practicing two effective methods of birth control
6. If female, must not be pregnant, plan to become pregnant, or nurse a child during the study and through 30 days after completion of the study
7. If male, must be surgically sterile or willing to practice two effective methods of birth control
8. Ability to understand and give informed consent

Exclusion Criteria:

1. Subjects with any evidence of respiratory infection including any signs or symptoms of either a lower respiratory infection (LRI) or upper respiratory infection (URI)
2. Known history of chronic pulmonary disease
3. Subjects who are being treated for fungal, viral, or bacterial pneumonia
4. Exposure to any investigational agent (defined as any agent not approved by the Food and Drug Administration [FDA]) within 30 days prior to the Screening Visit
5. Patients with a relapsed and/or refractory underlying hematologic malignancy
6. HSCT recipients who underwent ex vivo T-cell depletion of the graft, or a mismatched, or cord or haplo identical blood transplantation
7. HSCT recipients with active and/or chronic graft versus host disease
8. Patients on systemic corticosteroids (oral or intravenous)
9. Absolute neutrophil count (ANC) < 1,000 cells/mL
10. Clinically significant bacteremia or fungemia
11. Current smokers or subjects with any history of smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Forced Expiratory Volume in one Second (FEV1) | 3 weeks
  Evaluation of increasing doses of PUL-042 Inhalation Solution on FEV1

SECONDARY OUTCOMES:
Serum proteomics | 3 weeks
  Evalution of increasing doses of PUL-042 Inhalation Solution on serum proteomic profile

CONTACTS AND LOCATIONS:
Overall Officials: Roy F Chemaly, MD, MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No